CLINICAL TRIAL: NCT03782727
Title: Observational Study to Estimate the Proportion of Post-operative Infection Following Excision of Ulcerated Skin Tumours
Brief Title: ObservAtional Study to Investigate Surgical Site Infection in Ulcerated Skin Cancers
Acronym: OASIS
Status: Completed | Type: Observational
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: Cardiff University (Other); UK Dermatology Clinical Trials Network (Network)
Responsible Party: Principal Investigator, Rachel Abbott, Dermatology Consultant, Cardiff and Vale University Health Board
Other Study IDs: RD 17/DEC/7165
Record Dates: First submitted 2018-12-19; First posted 2018-12-20 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Skin Cancer
Keywords: skin cancer; surgery; ulcerated; infection
MeSH Terms: conditions — Skin Neoplasms; Ulcer; Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Participants enrolled to the study at University Hospital Cardiff will have swabs of ulcerated skin tumours taken and analysed in the Public Health Wales laboratory at the University of Wales, Cardiff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aim to recruit 311 participants to this study from three UK Dermatology departments. The investigators will invite people with suspected skin cancers whose lesions have a broken surface (also known as ulcerated) who will undergo surgery.

This study is being carried out because it is possible that patients with skin cancers with ulceration might be at greater risk of developing a wound infection after surgery. The aim of this study is to determine how many people with ulcerated skin cancers develop an infection of the wound after it has been surgically removed.

People with ulcerated skin cancers who will have surgery will be invited to participate in the study. If they agree, a member of the research team will explain the study and consent them to participate in the study. At the time of surgery, information will be collected about the participant, skin tumour and procedure. The participant will be given standardised advice regarding wound care and further care will be as per each centre's 'normal clinical care'. If participants are diagnosed with a wound infection then they will asked to take a 'wound selfie' and share the photo with the research team. The research team will contact the participant via a postal questionnaire which will be sent four weeks after the procedure to determine whether they had any concerns about post-operative infection and whether any action was taken.

Additionally, all participants at the University Hospital of Wales will have a surface swab taken from their ulcerated skin cancer and these will be analysed in the Public Health Wales laboratory at the University of Wales, Cardiff. The aim of this aspect of the study is to identify the most common bacteria in ulcerated tumours.

DETAILED DESCRIPTION:
Clinicians in the dermatology departments will identify eligible participants at the time of initial consultation. An information leaflet will be provided and details of the participants who are interested in participating will be forwarded to the research team to check eligibility prior to the procedure. Prior to the procedure relevant clinical information will be recorded in the Case Report Form (CRF) including demographic data, tumour site, tumour size, size of tumoural ulceration and type of wound closure. Histopathological data will be collected on tumour type when it is reported. Participants and clinicians will be asked whether they would agree for the patients to be randomised to no antibiotics, topical treatment eg. InadineTM dressings, a short course of antibiotics or a longer course of antibiotics in a future RCT. Following the procedure, information about whether oral antibiotics were prescribed will be recorded on a standardized CRF. All participants will be provided with the same information leaflet detailing standard post-operative advice and further care will be as per each centre's 'standard clinical care' which will also be recorded.

If participants are diagnosed with SSI they will be asked to take a photo of their wound on a camera phone and then to share the photo with the Cardiff University Centre for Trials Research (CTR) via email. Reeves et al. have described this practice as a 'wound selfie' and report that the term is readily understood. If participants are not able to take of photo of their wound then they will be invited to attend the department to have a photograph taken by medical photography. All participants will be sent a questionnaire by the research team four weeks following their procedure to enquire specifically whether the participant was diagnosed and treated for wound infection. These data will be collected by Cardiff University CTR who will co-ordinate the study.

Additionally, all participants at University Hospital of Wales will have a surface swab taken from their ulcerated skin tumour and these will be analysed in the Public Health Wales laboratory at the University of Wales, Cardiff. The aim of this aspect of the study is to identify the most common organisms that colonise ulcerated tumours. Previous studies have commented on growth from ulcerated tumours, however it is not clear if this was conducted in a research laboratory setting. This will help to guide antibiotic choice in a future randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1) at least 18 years old

Exclusion Criteria:

1. Evidence of wound infection at the time of the procedure
2. Skin tumour removal undertaken curettage or Mohs micrographic surgery
3. People without the capacity to consent for the study
4. People who are on systemic immunosuppressive treatment
5. People who are already taking oral antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People undergoing surgical excision of ulcerated skin cancer of any type at any body site in the dermatology departments at the University Hospital of Wales Cardiff; Churchill Hospital, Oxford and Queen Elizabeth Hospital, Birmingham.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Oxford University Hospitals NHS Foundation Trust, Oxford, England
  - Cardiff and Vale University Health Board, Cardiff, Wales
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Consented: Consecutive adult patients aged 18 years old or older who presented at either centre's outpatient department for an ulcerated skin cancer excision of any type in any body site were invited to participate.
Period: Overall Study
Arm/Group | Participants Consented
Started | 148
Completed | 116
Not Completed | 32
Not completed — Lost to Follow-up | 32

BASELINE CHARACTERISTICS:
Groups:
- Overall: Adult patients undergoing surgical excision of ulcerated skin cancer under local anaesthetic.
Arm/Group | Overall
Number analyzed (Participants) | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.1 (12.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 105
  Gender: Female | 41
  Gender: Missing data | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 148

OUTCOME MEASURES:

1. Primary Outcome: To Ascertain the Percentage of Surgical Site Infections Following Excision of Ulcerated Skin Tumours in Dermatology Departments.
Description: Percentage of participants with surgical site infection (SSI) identified by online/ postal questionnaire (Bluebelle Wound Healing Questionnaire) four weeks after surgery.
Time Frame: Four weeks after surgery.
Population: Proportion of participants with surgical site infection (SSI) identified by postal questionnaire (Bluebelle Wound Healing Questionnaire) four weeks after surgery (with score of 8 and above).
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Consented
Number analyzed (Participants) | 116
Participants | 35

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Participants Consented
All-Cause Mortality (participants affected / at risk) | 0/148
Serious Adverse Events (participants affected / at risk) | 0/148
Other Adverse Events (participants affected / at risk) | 0/148

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT03782727/Prot_SAP_000.pdf
  • Informed Consent Form: Consent form (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT03782727/ICF_001.pdf
  • Informed Consent Form: Patient Information leaflet (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT03782727/ICF_002.pdf